CLINICAL TRIAL: NCT03786029
Title: Comparison of Pre-emptive Ibuprofen, Acetaminophen, and Placebo Administration in Reducing Local Anesthesia Injection Pain and Post-operative Pain in Primary Tooth Extraction. A Clinical Study
Brief Title: Pre-emptive Analgesic Administration in Primary Tooth Extraction
Status: Completed | Phase: Phase 2 / Phase 3 | Type: Interventional
Sponsor: Tishreen University (Other)
Responsible Party: Principal Investigator, Nabih Raslan, Principal Investigator, Tishreen University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: Tishreen - Pre-emptive
Record Dates: First submitted 2018-12-15; First posted 2018-12-24 (Actual); Last update posted 2019-06-18 (Actual); Status verified 2019-06

CONDITIONS: Local Anesthesia; Tooth Extraction
Keywords: Pre-emptive administration; Analgesic; Tooth extraction
MeSH Terms: interventions — Acetaminophen; Ibuprofen

STUDY DESIGN:
Intervention Model Description: Blinded, randomized placebo-controlled trial, comparing three groups.
Who Masked: Participant, Investigator
Masking Description: The participant will be blinded, the drug administrator will be blinded too, and the investigator who will give the treatment and explain the pain scale to the participant and ask him\her to point to the face that fits the degree of his pain that associated with the drug administration will also be blinded.
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- A (Acetaminophen) (Experimental): 22 children will receive 320mg (10ml) 30 minutes before the local anesthesia injection.
  Interventions: Drug: Acetaminophen
- B (Placebo) (Placebo Comparator): 22 children will receive 10ml 30 minutes before the local anesthesia injection.
  Interventions: Drug: Placebo
- C (Ibuprofen) (Experimental): 22 children will receive 200mg (10ml) 30 minutes before the local anesthesia injection.
  Interventions: Drug: Ibuprofen

INTERVENTIONS:
Drug: Acetaminophen — Patients will receive 320mg (10ml) Acetaminophen (Strawberry flavour), wait for 30 minutes after the administration, then they will be given the local anesthesia injection. Then the child will be asked to point to the face that fits the degree of pain on the self-reporting pain scale WBFS immediately after the injection.
  The tooth will be extracted 10 minutes after the injection, then the child will be asked to record the degree of pain on the same scale immediately after the extraction.
  Pain will be re-evaluated 15 minutes after the extraction.
  The scale will be given to the parents in order to evaluate the post-extraction pain in 1 to 6 hours while the child is at home.
  Parents' satisfaction will be evaluated using Likert fifth scale.
  Other Names: A
  Arms: A (Acetaminophen)
Drug: Placebo — Patients will receive 10ml Strawberry Juice (placebo), wait for 30 minutes after the administration, then they will be given the local anesthesia injection. Then the child will be asked to point to the face that fits the degree of pain on the self-reporting pain scale WBFS immediately after the injection.
  The tooth will be extracted 10 minutes after the injection, then the child will be asked to record the degree of pain on the same scale immediately after the extraction.
  Pain will be re-evaluated 15 minutes after the extraction.
  The scale will be given to the parents in order to evaluate the post-extraction pain in 1 to 6 hours while the child is at home.
  Parents' satisfaction will be evaluated using Likert fifth scale.
  Other Names: B
  Arms: B (Placebo)
Drug: Ibuprofen — Patients will receive 200mg (10ml) of Ibuprofen (Strawberry flavour), wait for 30 minutes after the administration, then they will be given the local anesthesia injection. Then the child will be asked to point to the face that fits the degree of pain on the self-reporting pain scale WBFS immediately after the injection.
  The tooth will be extracted 10 minutes after the injection, then the child will be asked to record the degree of pain on the same scale immediately after the extraction.
  Pain will be re-evaluated 15 minutes after the extraction.
  The scale will be given to the parents in order to evaluate the post-extraction pain in 1 to 6 hours while the child is at home.
  Parents' satisfaction will be evaluated using Likert fifth scale.
  Other Names: C
  Arms: C (Ibuprofen)

SUMMARY:
Brief Summary:

Aims: The objective of the current study will be to compare the effectiveness of Ibuprofen, Acetaminophen, and Placebo on reducing injection pain and post-operative pain in primary tooth extraction, and to compare the parents' satisfaction.

Design: This will be a blinded, randomized placebo-controlled trial including sixty six cooperative children, aged 6-8 years old.

DETAILED DESCRIPTION:
Background and Aims: The pain could be a problem for the patients during the first few hours after the extraction because of both soft and hard tissues trauma during the operation, despite that the local anesthesia will last for a long time in most of the cases.

There are no enough studies that ensure the validity of giving any analgesic in reducing injection pain and post-operative pain in primary tooth extraction so far.

Design: This will be a blinded, randomized placebo-controlled trial including sixty six cooperative children, aged 6-8 years old, randomly assigned to one of three groups to receive one of the oral suspension drugs, that have the same colour and taste, via pre-calibrated medication bottles, which are identical, numbered and containing the same amount of pre-calibrated dosages, as per the following portions:

1. Acetaminophen syrup: 160mg/5ml
2. Placebo solution
3. Ibuprofen suspension: 100mg/5ml

ELIGIBILITY:
Inclusion Criteria:

1. Teeth with an abscess or infection exceeding one-third of the interradicular area (not exceeding the oral cavity) 2. Unrestorable decayed teeth. 3. Teeth with periapical / interradicular lesions.

-

Exclusion Criteria:

Teeth with advanced root resorption (a third of the root at least)

Ages: 6 Years to 8 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 66 (Actual)
Dates: Start 2019-04-01 (Actual); Primary Completion 2019-06-01 (Actual); Study Completion 2019-06-10 (Actual)

PRIMARY OUTCOMES:
Assessment pain related to the injection of the local anesthesia using WBFS. | 30-60 seconds after injection of the local anesthesia.
  The Wong-Baker Faces Pain Rating Scale (WBFS) is a pain scale that shows a series of faces ranging from a happy face at 0, or "no hurt", to a crying face at 10, which represents "hurts like the worst pain imaginable". Based on the faces and written descriptions, the patient chooses the face that best describes their level of pain.
  Immediately after the injection, the child will be asked to point to the face that fits the degree of pain on the self-reporting pain scale, WBFS.
Post operative pain assessment using WBFS. | 10 minutes - 6 hours after the extraction.
  After 10minutes from the injection and immediately after the extraction, the child will be asked to point to the face that fits the degree of pain on the same scale.
  Re-evaluate the pain after 15minutes from the extraction.
  The scale will be given to the parents to evaluate the pain post-extraction after an hour to 6 hours while the child is at home.

SECONDARY OUTCOMES:
Evaluate the parents' satisfaction using Likert fifth scale. | 6 hours after extraction.
  After the post-operation pain assessment is being done by the parents, the Likert fifth scale is used to determined the degree of parents satisfaction by choosing one of the following degrees: strongly agree, agree, neutral, disagree, strongly disagree.

CONTACTS AND LOCATIONS:
Overall Officials: Nabih Raslan, Dr, Study Chair — Tishreen University
Locations (1):
- Tishreen University, Latakia, Syria

IPD SHARING:
Plan to Share IPD: Undecided
Up to date, there is no decision about IPD sharing.

REFERENCES:
- [Background] Ashley PF, Parekh S, Moles DR, Anand P, MacDonald LC. Preoperative analgesics for additional pain relief in children and adolescents having dental treatment. Cochrane Database Syst Rev. 2016 Aug 8;2016(8):CD008392. doi: 10.1002/14651858.CD008392.pub3. PMID 27501304
- [Background] Pozos-Guillen A, Martinez-Rider R, Aguirre-Banuelos P, Perez-Urizar J. Pre-emptive analgesic effect of tramadol after mandibular third molar extraction: a pilot study. J Oral Maxillofac Surg. 2007 Jul;65(7):1315-20. doi: 10.1016/j.joms.2006.10.079. PMID 17577495
- [Background] Gazal G, Mackie IC. A comparison of paracetamol, ibuprofen or their combination for pain relief following extractions in children under general anaesthesia: a randomized controlled trial. Int J Paediatr Dent. 2007 May;17(3):169-77. doi: 10.1111/j.1365-263X.2006.00806.x. PMID 17397460
- [Background] Baygin O, Tuzuner T, Isik B, Kusgoz A, Tanriver M. Comparison of pre-emptive ibuprofen, paracetamol, and placebo administration in reducing post-operative pain in primary tooth extraction. Int J Paediatr Dent. 2011 Jul;21(4):306-13. doi: 10.1111/j.1365-263X.2011.01124.x. Epub 2011 Apr 6. PMID 21470320
- [Background] Ashkenazi M, Blumer S, Eli I. Post-operative pain and use of analgesic agents in children following intrasulcular anaesthesia and various operative procedures. Br Dent J. 2007 Mar 10;202(5):E13; discussion 276-7. doi: 10.1038/bdj.2007.81. Epub 2007 Feb 2. PMID 17273178
- [Background] Jurgens S, Warwick RS, Inglehearn PJ, Gooneratne DS. Pain relief for paediatric dental chair anaesthesia: current practice in a community dental clinic. Int J Paediatr Dent. 2003 Mar;13(2):93-7. doi: 10.1046/j.1365-263x.2003.00430.x. PMID 12605626
- [Background] Primosch RE, Nichols DL, Courts FJ. Comparison of preoperative ibuprofen, acetaminophen, and placebo administration on the parental report of postextraction pain in children. Pediatr Dent. 1995 May-Jun;17(3):187-91. PMID 7617493
- [Background] McGaw T, Raborn W, Grace M. Analgesics in pediatric dental surgery: relative efficacy of aluminum ibuprofen suspension and acetaminophen elixir. ASDC J Dent Child. 1987 Mar-Apr;54(2):106-9. PMID 3470325